CLINICAL TRIAL: NCT02521376
Title: A Phase 1, Open-Label, Multiple Dose Study to Evaluate the Pharmacokinetics of Entospletinib in Subjects With Normal and Impaired Hepatic Function
Brief Title: Pharmacokinetics of Entospletinib in Adults With Normal and Impaired Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-339-1631; 2016-003266-98 (EudraCT Number)
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms | interventions — 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Moderate Hepatic Impairment) (Experimental): Entospletinib administered twice daily on Days 1-4, and 1 morning dose only on Day 5.
  Interventions: Drug: Entospletinib
- Cohort 2 (Severe Hepatic Impairment) (Experimental): Entospletinib administered twice daily on Days 1-4, and 1 morning dose only on Day 5.
  Interventions: Drug: Entospletinib
- Cohort 3 (Mild Hepatic Impairment) (Experimental): Entospletinib administered twice daily on Days 1-4, and 1 morning dose only on Day 5.
  Interventions: Drug: Entospletinib

INTERVENTIONS:
Drug: Entospletinib — Entospletinib 100 mg tablet administered orally
  Other Names: GS-9973

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics of entospletinib (ENTO) and/or its metabolites (if applicable) in participants with impaired hepatic function (stratified by smoking status, as appropriate) relative to matched, healthy controls.

ELIGIBILITY:
Key Inclusion Criteria:

* Calculated body mass index from 18 to 40 kg/m^2
* Not pregnant
* Normal electrocardiogram
* Participants with impaired liver function must be sufficiently healthy based upon medical history and physical examination, vital signs, and screening laboratory evaluations.

Key Exclusion Criteria:

* Participation in another clinical study (current or within last 30 days)
* HIV, hepatitis B virus, or active hepatitis C virus infection

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (4):
  - Clinical Pharmacology of Miami, Inc. (CPMI), Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - The Texas Liver Institute, San Antonio, Texas
- APEX GmBH, Munich, Germany
- Auckland Clinical Studies, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States, New Zealand, and Germany. The first participant was screened on 16 November 2015. The last study visit occurred on 25 October 2017.
Pre-assignment Details: 102 participants were screened.
Groups:
- Severe Hepatic Impairment: Participants with severe hepatic impairment received entospletinib (ENTO) 100 mg tablet twice daily on Days 1-4, and 1 morning dose only on Day 5.
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment received ENTO 100 mg tablet twice daily on Days 1-4, and 1 morning dose only on Day 5.
- Mild Hepatic Impairment: Participants with mild hepatic impairment received ENTO 100 mg tablet twice daily on Days 1-4, and 1 morning dose only on Day 5.
- Healthy Control: Participants with normal hepatic function received ENTO 100 mg tablet twice daily on Days 1-4, and 1 morning dose only on Day 5.
Period: Overall Study
Arm/Group | Severe Hepatic Impairment | Moderate Hepatic Impairment | Mild Hepatic Impairment | Healthy Control
Started | 8 | 18 | 10 | 20
Completed | 7 | 18 | 10 | 20
Not Completed | 1 | 0 | 0 | 0
Not completed — Enrolled, But Not Treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe Hepatic Impairment | Moderate Hepatic Impairment | Mild Hepatic Impairment | Healthy Control | Total
Number analyzed (Participants) | 7 | 18 | 10 | 20 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (10.6) | 59 (8.5) | 58 (11.4) | 56 (9.3) | 57 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5 | 5 | 15
  Male | 6 | 14 | 5 | 15 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 3 | 9 | 20
  Not Hispanic or Latino | 4 | 13 | 7 | 11 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2 | 4
  White | 7 | 17 | 9 | 17 | 50
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 1 | 0 | 1 | 0 | 2
  United States | 5 | 17 | 8 | 19 | 49
  Germany | 1 | 1 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of ENTO
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60, 72, 84, and 96 hours postdose on Day 5
Population: Participants in the PK Analysis Set (all enrolled participants who received at least one dose of ENTO and had at least one evaluable PK concentration data value reported by the PK lab) with available data were analyzed. Healthy control participants may participate in more than one cohorts.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Cohort 1: Moderate Hepatic Impairment Smoking: Participants with moderate hepatic impairment who are smokers received ENTO 100 mg tablet twice daily on Days 1-4, and 1 morning dose only on Day 5.
- Cohort 1: Moderate Hepatic Impairment Non-smoking: Participants with moderate hepatic impairment who are non-smokers received ENTO 100 mg tablet twice daily on Days 1-4, and 1 morning dose only on Day 5.
- Cohort 1: Healthy Control Matched to Smoking: Participants with normal hepatic function who are smokers received ENTO 100 mg tablet twice daily on Days 1-4, and 1 morning dose only on Day 5.
- Cohort 1: Healthy Control Matched to Non-smoking: Participants with normal hepatic function who are non-smokers received ENTO 100 mg tablet twice daily on Days 1-4, and 1 morning dose only on Day 5.
- Cohort 2: Severe Hepatic Impairment: Participants with severe hepatic impairment received ENTO 100 mg tablet twice daily on Days 1-4, and 1 morning dose only on Day 5.
- Cohort 2: Healthy Control; Cohort 3: Healthy Control: Participants with normal hepatic function received ENTO 100 mg tablet twice daily on Days 1-4, and 1 morning dose only on Day 5.
- Cohort 3: Mild Hepatic Impairment: Participants with mild hepatic impairment received ENTO 100 mg tablet twice daily on Days 1-4, and 1 morning dose only on Day 5.
Arm/Group | Cohort 1: Moderate Hepatic Impairment Smoking | Cohort 1: Moderate Hepatic Impairment Non-smoking | Cohort 1: Healthy Control Matched to Smoking | Cohort 1: Healthy Control Matched to Non-smoking | Cohort 2: Severe Hepatic Impairment | Cohort 2: Healthy Control | Cohort 3: Mild Hepatic Impairment | Cohort 3: Healthy Control
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 7 | 7 | 10 | 10
h*ng/mL | 1788.9 (771.30) | 7490.0 (3805.03) | 4081.5 (2464.77) | 3318.0 (1788.90) | 7036.0 (2814.95) | 3402.7 (1771.79) | 4071.9 (913.47) | 4123.0 (1874.33)
Statistical Analysis 1: Comparison: Cohort 1: Moderate Hepatic Impairment Smoking vs Cohort 1: Healthy Control Matched to Smoking; Test type: Other; Geometric Mean Ratio (GMR) = 43.69, 90% CI 2-sided [24.59 to 77.62]
Statistical Analysis 2: Comparison: Cohort 1: Moderate Hepatic Impairment Non-smoking vs Cohort 1: Healthy Control Matched to Non-smoking; Test type: Other; GMR = 233.63, 90% CI 2-sided [141.85 to 384.79]
Statistical Analysis 3: Comparison: Cohort 2: Severe Hepatic Impairment vs Cohort 2: Healthy Control; Test type: Other; GMR = 219.20, 90% CI 2-sided [139.74 to 343.84]
Statistical Analysis 4: Comparison: Cohort 3: Mild Hepatic Impairment vs Cohort 3: Healthy Control; Test type: Other; GMR = 108.50, 90% CI 2-sided [77.20 to 152.48]

2. Primary Outcome: Pharmacokinetic (PK) Parameter: Cmax of ENTO
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60, 72, 84, and 96 hours postdose on Day 5
Population: Participants in the PK Analysis Set with available data were analyzed. Healthy control participants may participate in more than one cohorts.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Moderate Hepatic Impairment Smoking | Cohort 1: Moderate Hepatic Impairment Non-smoking | Cohort 1: Healthy Control Matched to Smoking | Cohort 1: Healthy Control Matched to Non-smoking | Cohort 2: Severe Hepatic Impairment | Cohort 2: Healthy Control | Cohort 3: Mild Hepatic Impairment | Cohort 3: Healthy Control
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 7 | 7 | 10 | 10
ng/mL | 313.1 (122.39) | 1007.3 (480.63) | 582.3 (326.04) | 497.4 (292.67) | 837.7 (326.52) | 521.1 (280.65) | 569.8 (166.56) | 590.5 (326.08)
Statistical Analysis 1: Comparison: Cohort 1: Moderate Hepatic Impairment Smoking vs Cohort 1: Healthy Control Matched to Smoking; Test type: Other; GMR = 55.71, 90% CI 2-sided [34.70 to 89.42]
Statistical Analysis 2: Comparison: Cohort 1: Moderate Hepatic Impairment Non-smoking vs Cohort 1: Healthy Control Matched to Non-smoking; Test type: Other; GMR = 211.94, 90% CI 2-sided [132.49 to 339.03]
Statistical Analysis 3: Comparison: Cohort 2: Severe Hepatic Impairment vs Cohort 2: Healthy Control; Test type: Other; GMR = 171.33, 90% CI 2-sided [108.17 to 271.37]
Statistical Analysis 4: Comparison: Cohort 3: Mild Hepatic Impairment vs Cohort 3: Healthy Control; Test type: Other; GMR = 107.35, 90% CI 2-sided [72.71 to 158.51]

3. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as events that meet one of the following criteria:
  * Any adverse events (AEs) with onset date of on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug or
  * Any AEs leading to premature discontinuation of study drug.
Time Frame: Baseline up to Day 9 plus 30 days
Population: Safety Analysis Set included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Severe Hepatic Impairment | Moderate Hepatic Impairment | Mild Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 7 | 18 | 10 | 20
percentage of participants | 14.3 | 22.3 | 30.0 | 30.0

4. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each subject.
Time Frame: Baseline up to Day 9 plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Severe Hepatic Impairment | Moderate Hepatic Impairment | Mild Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 7 | 18 | 10 | 20
percentage of participants | 100.0 | 88.9 | 60.0 | 50.0

ADVERSE EVENTS:
Time Frame: First dose date up to Day 9 plus 30 days
Description: Safety Analysis Set included all randomized participants who received at least one dose of study drug.
Arm/Group | Severe Hepatic Impairment | Moderate Hepatic Impairment | Mild Hepatic Impairment | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/18 | 0/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/18 | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 1/7 | 4/18 | 3/10 | 6/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Hepatic Impairment (N=7) | Moderate Hepatic Impairment (N=18) | Mild Hepatic Impairment (N=10) | Healthy Control (N=20)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Infected bite (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 4
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (6):
  • Study Protocol: Original (2015-07-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT02521376/Prot_000.pdf
  • Study Protocol: Amendment 1 (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT02521376/Prot_001.pdf
  • Study Protocol: Amendment 2 (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT02521376/Prot_002.pdf
  • Study Protocol: Amendment 3 (2016-08-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT02521376/Prot_003.pdf
  • Study Protocol: Amendment 4 (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT02521376/Prot_004.pdf
  • Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT02521376/SAP_005.pdf